CLINICAL TRIAL: NCT05132673
Title: Cardiac Autonomic Dysfunction in Childhood Cancer Survivors
Status: Suspended | Type: Observational
Why Stopped: Placing the study on HOLD to recruitment to minimize the number of recruitment emails potential participants will receive. Our goal is to resubmit the grant that will fund this protocol as part of the next grant submission cycle in February 2023.
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: WEARIT; NCI-2022-00145 (Registry Identifier: NCI)
Record Dates: First submitted 2021-10-06; First posted 2021-11-24 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Autonomic Dysfunction; Childhood Cancer
Keywords: childhood cancer survivors; cardiac
MeSH Terms: conditions — Primary Dysautonomias; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants: Those who meet the Eligibility Criteria will be asked to complete online questionnaires and wear a device on your wrist for two weeks that measures your heart rate, physical activity, and sleep. A WHOOP® wrist monitor and charging equipment will be used.

SUMMARY:
This study is being done to evaluate heart rate activity and sleep patterns, among participants in the Long-Term Follow-Up (LTFU) study.

Primary Objective

Using mobile health (mHealth) technologies in a large and well-characterized cohort of childhood cancer survivors, our primary objective is to understand the magnitude of increased risk of cardiac autonomic dysfunction by (a) comparing prevalence rates among survivors and siblings, and (b) determining the prevalence within specific subgroups of childhood cancer survivors defined by race, sex, cancer type and treatment exposures, and type and severity of chronic health conditions.

Secondary Objectives

Among long-term (≥5 years) survivors of childhood cancer (a) identify demographic, disease, treatment and cognitive-behavioral factors associated with an increased risk of cardiac autonomic dysfunction, (b) develop and validate risk prediction models for future clinical use in identifying individuals who may benefit from targeted interventions, and (c) investigate associations between dysfunction and perceived well-being.

DETAILED DESCRIPTION:
Potential participants will be recruited by email and phone. Survivors who wish to participate will complete an online consent form and then a series of short questionnaires to determine study eligibility. This data collection will take place in DatStat Connect, which is the online consenting and data collection tool utilized for the CCSS. Consented/enrolled SJLIFE participants will receive a link via email to complete surveys related to autonomic functioning and current medical concerns and asked to schedule delivery of a WHOOP® strap prior kit prior to scheduling a device setup session with a team member. The kit will include the WHOOP® strap, brief instructions for setup, and prepaid return mailing materials. The WHOOP® strap will be shipped to the participant and each participant will complete a training session and app installation, if needed, and instructions regarding during of wear (two weeks)

ELIGIBILITY:
Inclusion Criteria:

* Enrollment on the CCSS protocol.
* 18 years or older.
* Has a smartphone and is willing to download the WHOOP® app for the duration of study participation.
* Reports no history of allergic reaction (e.g., rash) to fitness monitoring wearables.

Exclusion Criteria:

* Unable to independently provide informed consent.
* Visual impairment that prevents participant from engaging with study materials.
* Unable to read or understand study materials in English.
* Mailing address outside the United States.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Those who meet the eligibility criteria
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Heart rate variability | Measured over a 24 hour period
  Standard deviation of NN (normal to normal RR) intervals (SDNN)

SECONDARY OUTCOMES:
Autonomic Symptoms | Assessed at baseline
  Self-reported autonomic symptoms via the COMPASS31
Perceived health | Assessed at baseline
  Self-reported perceived health via Medical Outcomes Study 36-Item Short-Form Health Survey (SF-36)
Perceived stress | Assessed at baseline
  Cohen's Perceived Stress Scale, Minimum value = 0, Maximum value = 40, Higher scores mean a worse outcome
Cognitive status | Assessed at baseline
  Childhood Cancer Survivor Study Neurocognitive Questionnaire, Minimum Value = 33, Maximum value = 99, Higher scores mean a worse outcome
Sleep Onset | Measured over 2 weeks
  Sleep hygiene will be measured via wearable sleep tracker. Sleep onset will be measured in minutes.
Wake Onset | Measured daily over 2 weeks
  Sleep hygiene will be measured via wearable sleep tracker. Wake onset will be measured in minutes.
Sleep efficiency | Measured daily over 2 weeks
  Sleep hygiene will be measured via wearable sleep tracker. Sleep efficient will be measured by dividing the minutes asleep by the total minutes in bed.
Physical activity duration | Measured daily over 2 weeks
  Intensity and duration of daily activity will be measured via wearable activity tracker. Activity duration will be measured in minutes.
Workout strain | Measured daily over 2 weeks
  Intensity and duration of daily activity will be measured via wearable activity tracker. Workout strain will be calculated by the duration of time in personal heart rate zones, established from maximum heart rate.
Maximum heart rate | Measured daily over 2 weeks
  Intensity and duration of daily activity will be measured via wearable activity tracker. Maximum heart rate will be calculated by subtracting age from 220 and is measured in beats per minute.
Average heart rate | Measured daily over 2 weeks
  Intensity and duration of daily activity will be measured via wearable activity tracker. Average heart rate will be calculated as number of beats per minute.

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten Ness, PhD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols